CLINICAL TRIAL: NCT03413969
Title: Building Physician Resiliency Through CREATION Health: A Research Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been terminated due to recruitment challenges in targeted area.
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1090321
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Burnout; Stress; Well-being
MeSH Terms: conditions — Burnout, Psychological | interventions — Facility Design and Construction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Intervention (Experimental): The study subjects will be recruited for approximately six weeks prior to the projected start date. The participants will attend the two-day weekend retreat. Follow-up assessments will be administered three months and six months after the retreat. The investigators will analyze the data and complete the study one month after the final assessment is administered.
  Interventions: Behavioral: CREATION

INTERVENTIONS:
Behavioral: CREATION — The physician-oriented intervention will consist of a two-day weekend retreat that focuses on the application of CREATION Health principles in order to reduce burnout and perceived stress and improve well-being and empathy. There will be one four-hour session about each of the following CREATION Health principles: Choice, Trust, Interpersonal Relationships, and Outlook.

SUMMARY:
The purpose of this study is to determine whether a standardized application of a physician-oriented CREATION Health curriculum is associated with reductions in burnout and perceived stress and improvements in well-being and empathy

DETAILED DESCRIPTION:
This is a prospective, non-randomized study of a convenience sample of Centura Health physicians.This study will not include any drugs or devices. The physician-oriented intervention will consist of a two-day weekend retreat that focuses on the application of CREATION Health principles in order to reduce burnout and perceived stress and improve well-being and empathy. There will be one four-hour session about each of the following CREATION Health principles: Choice, Trust, Interpersonal Relationships, and Outlook.

ELIGIBILITY:
Inclusion Criteria:

* Physician employed by Centura Health or credentialed physician with privileges at Centura Health
* Adult ≥ 18 years old
* English language proficiency
* Able to provide informed consent
* Resides in the Denver, Colorado area
* Willing to commit to the timeline of the study

Exclusion Criteria:

* Plans to reside outside of the Denver, Colorado area within the 8 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory - Human Services Survey | 12 Months
  The Emotional Exhaustion subscale scores range from 0 to 54. Higher scores indicate worse outcomes. The Depersonalization subscale scores range from 0 to 30. Higher scores indicate worst outcomes. The Personal Accomplishment subscale scores range from 0 to 48. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Well-Being Item | 12 Months
  The following question will be asked to assess well-being: "How satisfied are you with your life as a whole?" The scores range from 0 to 10. Higher scores indicate better outcomes.

OTHER OUTCOMES:
Perceived Stress Scale | 12 Months
  The Perceived Stress Scale will be used to measure perceived stress. The scores range from 0 to 40. Higher scores indicate worse outcomes.
Jefferson Scale of Empathy | 12 Months
  The Jefferson Scale of Empathy will be used to assess empathy. The scores range from 0 to 140. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Terry, Principal Investigator — Center for CREATION Health Research
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shanafelt TD, Boone S, Tan L, Dyrbye LN, Sotile W, Satele D, West CP, Sloan J, Oreskovich MR. Burnout and satisfaction with work-life balance among US physicians relative to the general US population. Arch Intern Med. 2012 Oct 8;172(18):1377-85. doi: 10.1001/archinternmed.2012.3199. PMID 22911330
- [Background] Maslach C, Jackson SE, Leiter MP. Maslach Burnout Inventory manual. 3rd ed. Palo Alto, CA: Consulting Psychologists Press; 1996.
- [Background] Shanafelt TD, Noseworthy JH. Executive Leadership and Physician Well-being: Nine Organizational Strategies to Promote Engagement and Reduce Burnout. Mayo Clin Proc. 2017 Jan;92(1):129-146. doi: 10.1016/j.mayocp.2016.10.004. Epub 2016 Nov 18. PMID 27871627
- [Background] Shanafelt TD, Sloan JA, Habermann TM. The well-being of physicians. Am J Med. 2003 Apr 15;114(6):513-9. doi: 10.1016/s0002-9343(03)00117-7. No abstract available. PMID 12727590
- [Background] Wallace JE, Lemaire JB, Ghali WA. Physician wellness: a missing quality indicator. Lancet. 2009 Nov 14;374(9702):1714-21. doi: 10.1016/S0140-6736(09)61424-0. PMID 19914516
- [Background] O'Connor PG, Spickard A Jr. Physician impairment by substance abuse. Med Clin North Am. 1997 Jul;81(4):1037-52. doi: 10.1016/s0025-7125(05)70562-9. PMID 9222267
- [Background] Spickard A Jr, Gabbe SG, Christensen JF. Mid-career burnout in generalist and specialist physicians. JAMA. 2002 Sep 25;288(12):1447-50. doi: 10.1001/jama.288.12.1447. No abstract available. PMID 12243624
- [Background] Thomas NK. Resident burnout. JAMA. 2004 Dec 15;292(23):2880-9. doi: 10.1001/jama.292.23.2880. PMID 15598920
- [Background] Crane M. Why burned-out doctors get sued more often. Med Econ. 1998 May 26;75(10):210-2, 215-8. No abstract available. PMID 10179678
- [Background] Haas JS, Cook EF, Puopolo AL, Burstin HR, Cleary PD, Brennan TA. Is the professional satisfaction of general internists associated with patient satisfaction? J Gen Intern Med. 2000 Feb;15(2):122-8. doi: 10.1046/j.1525-1497.2000.02219.x. PMID 10672116
- [Background] Shanafelt TD, West C, Zhao X, Novotny P, Kolars J, Habermann T, Sloan J. Relationship between increased personal well-being and enhanced empathy among internal medicine residents. J Gen Intern Med. 2005 Jul;20(7):559-64. doi: 10.1111/j.1525-1497.2005.0108.x. PMID 16050855
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] West CP, Dyrbye LN, Erwin PJ, Shanafelt TD. Interventions to prevent and reduce physician burnout: a systematic review and meta-analysis. Lancet. 2016 Nov 5;388(10057):2272-2281. doi: 10.1016/S0140-6736(16)31279-X. Epub 2016 Sep 28. PMID 27692469
- [Background] Fujimori M, Oba A, Koike M, Okamura M, Akizuki N, Kamiya M, Akechi T, Sakano Y, Uchitomi Y. Communication skills training for Japanese oncologists on how to break bad news. J Cancer Educ. 2003 Winter;18(4):194-201. doi: 10.1207/s15430154jce1804_6. PMID 14766329
- [Background] Fujimori M, Shirai Y, Asai M, Akizuki N, Katsumata N, Kubota K, Uchitomi Y. Development and preliminary evaluation of communication skills training program for oncologists based on patient preferences for communicating bad news. Palliat Support Care. 2014 Oct;12(5):379-86. doi: 10.1017/S147895151300031X. Epub 2013 Nov 4. PMID 24182602
- [Background] Goodman MJ, Schorling JB. A mindfulness course decreases burnout and improves well-being among healthcare providers. Int J Psychiatry Med. 2012;43(2):119-28. doi: 10.2190/PM.43.2.b. PMID 22849035
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Background] Ospina-Kammerer V, Figley CR. An evaluation of the Respiratory One Method (ROM) in reducing emotional exhaustion among family physician residents. Int J Emerg Ment Health. 2003 Winter;5(1):29-32. PMID 12722487
- [Background] Rosdahl JA, Kingsolver KO. Mindfulness training to increase resilience and decrease stress and burnout in ophthalmology residents: A pilot study. Invest Ophthalmol Vis Sci. 2014;55(13):5579.
- [Background] Winefield H, Farmer E, Denson L. Work stress management for women general practitioners: An evaluation. Psychol Health Med. 1998;3(2):163-170.
- [Background] Dunn PM, Arnetz BB, Christensen JF, Homer L. Meeting the imperative to improve physician well-being: assessment of an innovative program. J Gen Intern Med. 2007 Nov;22(11):1544-52. doi: 10.1007/s11606-007-0363-5. Epub 2007 Sep 22. PMID 17891503
- [Background] International Wellbeing Group. Personal Wellbeing Index: 5th edition. Melbourne: Australian Centre on Quality of Life, Deakin University; 2013.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cohen S, Williamson G. Psychological stress in a probability sample of the United States. In: Spacapan S, Oskamp S, eds. The social psychology of health. Newbury Park, CA: Sage; 1988:31-67.
- [Background] Hojat M, Mangione S, Nasca T, et al. The Jefferson Scale of Physician Empathy: Development and Preliminary Psychometric Data. Educ Psychol Meas. 2001; 61(2):349-365.